CLINICAL TRIAL: NCT00198341
Title: Multicentric Randomized Phase III Study of Post-Surgical NSCLC Follow-up
Brief Title: Post-Surgical Non-Small Cell Lung Cancer (NSCLC) Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0302
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Post-surgical Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (2):
- 1 (Experimental): Radiological arm (Clinical Visit + X-Ray Chest)
  Interventions: Procedure: Radiological Arm
- 2 (Experimental): Scan ARM : Clinical Visit + X-Ray Chest + CT-Scan + Fibroscopy (for squamous type)
  Interventions: Procedure: Scannographic arm

INTERVENTIONS:
Procedure: Radiological Arm — Clinical Visit + X-Ray Chest
  Arms: 1
Procedure: Scannographic arm — Clinical visit + X-Ray Chest + CT-Scan + Fibroscopy (for squamous cell)
  Arms: 2

SUMMARY:
The follow-up of patients operated on for lung cancer is heterogeneous. An intensive follow-up including routine clinic visits, chest X-rays, chest computed tomography (CT) scans and fiberoptic bronchoscopies might detect more small, potentially curable, recurrences and second cancers. However, as it appears in the American Society of Clinical Oncology (ASCO) recommendations, a large randomized study is necessary to evaluate the survival impact of such a follow-up strategy. This is the main objective of this IFCT-0302 study, which is a large randomized controlled study conducted in France comparing this intensive follow-up to a follow-up with only routine clinic visits and chest X-rays.

ELIGIBILITY:
Inclusion Criteria:

* completely resected stage I, II, IIIa, and T4 due to satellite tumor nodule(s) N0-2 NSCLC

Exclusion Criteria:

* stage IIIb to IV NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1775 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Compare overall survival for each arm | 6-month

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Westeel, Pr, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (7):
- France (7):
  - Centre Hospitalier - Pneumologie, Belfort
  - CHU Besancon - Pneumologie, Besançon
  - Centre F. Baclesse, Caen
  - CHU - Pneumologie, Caen
  - CHU Grenoble - pneumologie, Grenoble
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - CHU Lyautey - Pneumologie, Strasbourg

REFERENCES:
- [Background] Westeel V, Lebitasy MP, Mercier M, Girard P, Barlesi F, Blanchon F, Tredaniel J, Bonnette P, Woronoff-Lemsi MC, Breton JL, Azarian R, Falcoz PE, Friard S, Geriniere L, Laporte S, Lemarie E, Quoix E, Zalcman G, Guigay J, Morin F, Milleron B, Depierre A; Intergroupe Francophone de Cancerologie Thoracique (IFCT). [IFCT-0302 trial: randomised study comparing two follow-up schedules in completely resected non-small cell lung cancer]. Rev Mal Respir. 2007 May;24(5):645-52. doi: 10.1016/s0761-8425(07)91135-3. French. PMID 17519819
- [Derived] Westeel V, Foucher P, Scherpereel A, Domas J, Girard P, Tredaniel J, Wislez M, Dumont P, Quoix E, Raffy O, Braun D, Derollez M, Goupil F, Hermann J, Devin E, Barbieux H, Pichon E, Debieuvre D, Ozenne G, Muir JF, Dehette S, Virally J, Grivaux M, Lebargy F, Souquet PJ, Freijat FA, Girard N, Courau E, Azarian R, Farny M, Duhamel JP, Langlais A, Morin F, Milleron B, Zalcman G, Barlesi F. Chest CT scan plus x-ray versus chest x-ray for the follow-up of completely resected non-small-cell lung cancer (IFCT-0302): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2022 Sep;23(9):1180-1188. doi: 10.1016/S1470-2045(22)00451-X. Epub 2022 Aug 11. PMID 35964621
- See also: official IFCT website — http://www.ifct.fr